CLINICAL TRIAL: NCT04806178
Title: Systemic Immunological Response of Bladder Cancer Patients Under Bacillus Calmette Guérin Treatment
Brief Title: Immunological Response of Bladder Cancer Patients Under BCG
Acronym: IMMUNOBCG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other); Pontifical University Catholic of Campinas (Other)
Responsible Party: Principal Investigator, Leonardo Oliveira Reis, Professor Livre Docente, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCG IMMUNO Bladder
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer; Bacillus Calmette-Guerin
Keywords: BCG; Bladder cancer; Immunotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG intradermal vaccine (Active Comparator): Intradermal BCG Group (n=16): 0.1 ml of lyophilized, live, and attenuated BCG intradermal vaccine, containing between 2 and 8 x 1.000.000 C.F.U in a single dose.
  Interventions: Biological: Bacillus Calmette Guerin
- Placebo (Placebo Comparator): Placebo group (n = 16): 0.9% saline solution in the same volume as BCG vaccine in a single dose.
  Interventions: Other: PLACEBO

INTERVENTIONS:
Biological: Bacillus Calmette Guerin — 0.1 ml of lyophilized, live, and attenuated BCG intradermal vaccine, containing between 2 and 8 x 1.000.000 C.F.U in a single dose.
  Other Names: BCG
  Arms: BCG intradermal vaccine
Other: PLACEBO — 0.1 ml 0.9% saline in the same volume as the BCG vaccine in a single dose.
  Arms: Placebo

SUMMARY:
Bladder cancer (BC) is one of the most common cancers worldwide and the most successful example of vaccine in cancer treatment, representing an efficient model for studying the importance of systemic and local immune mechanisms. Despite being the standard of treatment for the last 40 years, the exact mode of action of immunotherapy with the bacillus Calmette-Guérin (BCG) is still poorly defined. In a mechanistic study, the investigators intend to prospectively investigate immunological signatures, including immune-checkpoints, pre and post-treatment in patients with BC, and correlate the cytokines of the immune by-product and BCG administration pathway to understand the independent contributions of BCG priming (prior exposure to BCG) and crosstalk immunotherapy between tumor profiles and immune response of the patient. The proposed research strategy is justified by the need to identify subsets of patients who better respond to an intervention, or to predict why new immunotherapies and drugs may be successful or failed in clinical trials.

DETAILED DESCRIPTION:
Recognizing patient-to-patient variability, key data scarcity, and insight into traditional reductionist therapy, the BCG model offers exceptionally compelling opportunities to understand how immune system behavior in health and disease emerges from local, systemic, genetic, epigenetic, cellular, and environmental modulating factors.

The application seeks to change the current clinical practice and research paradigms, by using new theoretical concepts, challenging bladder cancer patients with a highly effective, safe, and affordable immunotherapy, the gold standard in the last 40 years of NMIBC, and in light of new concepts and methodologies brought by the paradigm of immune-checkpoint inhibitors that justified the Nobel Prize in Physiology or Medicine in 2018.

The current proposal has the potential to impact the prognosis and identification of those who are unlikely to respond to immune-checkpoint inhibitors, scenarios in which important unanswered questions remain, particularly as this class of agents advances along the spectrum of non-metastatic disease.

In a mechanistic approach, patients diagnosed with NMIBC and with the indication for intravesical BCG treatment will be randomized to placebo versus a priming intradermic BCG 14 days before the intravesical treatment and followed up to 180 days.

The investigators will define important clinical paradigms:

1. The role of the priming effect on the immune system and better understanding of BCG immunotherapy, with a clear potential for improvement of bladder cancer treatment in NMIBC and MIBC scenarios;
2. The potential of BCG, a widely used vaccine, to improve or impair the results of new immunotherapies, given its long-lasting effect;
3. Rational to develop future treatment associations of BCG and immune-checkpoints. \

Under the new immunological concepts, a better understanding of tumor-associated immune responses in BC patients could provide more informed clinical decisions and treatment optimization.

Considering the growing need of assessing the value of treatment at the expense of cost, part of our proposal strategy is to limit financial toxicity as an important issue in cancer treatment and new immunotherapies.

ELIGIBILITY:
Inclusion Criteria:

* NMIBC with the indication for intravesical BCG treatment;

Exclusion Criteria:

* Previous BCG treatment;
* Muscle invasive tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Flow Cytometry | Day 0
  Cellular Immune Response
Flow Cytometry | Day 14
  Cellular Immune Response
Flow Cytometry | Day 21
  Cellular Immune Response
Flow Cytometry | Day 35
  Cellular Immune Response
Flow Cytometry | Day 49
  Cellular Immune Response
Flow Cytometry | Day 180
  Cellular Immune Response

SECONDARY OUTCOMES:
Adverse Effects and Change from Baseline Voiding Symptoms | Day 21
  American Urological Association Symptom Score Questionnaire - minimum 0 and maximum 35, higher scores mean a worse outcome.
Adverse Effects and Change from Baseline Voiding Symptoms | Day 35
  American Urological Association Symptom Score Questionnaire - minimum 0 and maximum 35, higher scores mean a worse outcome.
Adverse Effects and Change from Baseline Voiding Symptoms | Day 49
  American Urological Association Symptom Score Questionnaire - minimum 0 and maximum 35, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo O Reis, MD, PhD, Principal Investigator — University of Campinas
Locations (2):
- Brazil (2):
  - Pontifical Catholic University of Campinas Hospital, Campinas, São Paulo
  - Hospital das Clínicas Unicamp, Campinas, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ji N, Mukherjee N, Morales EE, Tomasini ME, Hurez V, Curiel TJ, Abate G, Hoft DF, Zhao XR, Gelfond J, Maiti S, Cooper LJN, Svatek RS. Percutaneous BCG enhances innate effector antitumor cytotoxicity during treatment of bladder cancer: a translational clinical trial. Oncoimmunology. 2019 May 25;8(8):1614857. doi: 10.1080/2162402X.2019.1614857. eCollection 2019. PMID 31413921
- [Background] van Puffelen JH, Keating ST, Oosterwijk E, van der Heijden AG, Netea MG, Joosten LAB, Vermeulen SH. Trained immunity as a molecular mechanism for BCG immunotherapy in bladder cancer. Nat Rev Urol. 2020 Sep;17(9):513-525. doi: 10.1038/s41585-020-0346-4. Epub 2020 Jul 16. PMID 32678343